CLINICAL TRIAL: NCT05911568
Title: Treatment With Endovascular Intervention for STroke Patients With Existing Disability
Acronym: TESTED
Status: Recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of California, Los Angeles (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Eva A. Mistry, Assistant Professor, University of Cincinnati
Other Study IDs: 2023-0299
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Practice Management, Medical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients with moderate-to-severe pre-stroke disability: Patients with pre-stroke modified Rankin scale score 3 or 4, presenting with a anterior circulation large vessel occlusion stroke within 24 hours of last known well
  Interventions: Procedure: Endovascular Stroke Treatment; Other: Medical Management

INTERVENTIONS:
Procedure: Endovascular Stroke Treatment — Patients who receive endovascular stroke treatment when they are admitted into the hospital, as determined by their clinical care team. Endovascular stroke treatment consist of catheter-based treatment for the blood clot causing the acute ischemic stroke
Other: Medical Management — Patients who receive MMM when they are admitted into the hospital, as determined by their clinical care team. MMM may involve any combination of the following: intravenous thrombolysis, antiplatelets, anti-hypertensives, cholesterol-lowering medications, and rehabilitative care. Specifically, this treatment does not involve endovascular stroke treatment.

SUMMARY:
TESTED will compare the risks and benefits of endovascular thrombectomy (EVT) to medical management (no EVT) in ischemic stroke patients who have a blockage in one of the large blood vessels in the brain and have a moderate-to-severe disability prior to their stroke.

DETAILED DESCRIPTION:
People with disabilities can suffer acute ischemic stroke (AIS). Endovascular clot removal is a breakthrough therapy for large vessel occlusion (LVO) AIS. Pre-stroke disabled patients were excluded from pivotal EVT stroke trials, so whether EVT is effective for those with pre-stroke disability is not known. As a result, two competing, widely-practiced, treatment paradigms have emerged based on individual practitioners' extrapolation of EVT benefits and safety from patients without a pre-stroke disability to those with disability: 1) Multimodal Medical Management (MMM; using intravenous thrombolysis, antiplatelets, anti-hypertensives, cholesterol lowering medications, and other rehabilitative measures, as indicated) without EVT, and 2) EVT with the background of MMM.

TESTED will enroll patients with LVO-AIS who have a pre-existing disability, defined as pre-stroke modified Rankin score (mRS) 3 and 4, at 12 geographically distinct comprehensive stroke centers serving diverse race-ethnic and socioeconomic populations. The central objective of TESTED is to determine the comparative effectiveness and safety of these two different practice paradigms.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years)
2. Moderate-to-severe pre-stroke functional disability, defined as mRS 3-4, for at least 3 months prior to stroke onset
3. Presenting to study hospital within 24 hours of last known well time
4. Diagnosis of acute ischemic stroke
5. Intracranial causative occlusion of the internal carotid artery or the M1 or dominant M2 segments of the middle cerebral artery visualized on the baseline CT(or MR) angiogram
6. Presenting CT Alberta Stroke Program Early CT (ASPECT) score ≥3 or MRI ASPECT score ≥4
7. Presenting NIH Stroke Scale score ≥6
8. Informed consent from patient if competent or from legally authorized representative

Exclusion Criteria:

1. Known diagnosis of a terminal cancer or terminal illness at the time of stroke
2. Assessment of pre-stroke functional status cannot be performed during the hospital stay
3. Pre-stroke disability deemed temporary in the investigator's opinion (for example, recovering from a general medical illness or traumatic bodily injury)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients who have a blockage in one of the large blood vessels in the brain and have a moderate-to-severe disability prior to their stroke. They will be consented up to 72 hours after stroke onset in the acute hospitalization setting.
Sampling Method: Non-Probability Sample
Enrollment: 1060 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) | 90 (±14) days after treatment initiation
  Score of 0-3, 4, 5 or 6 on the modified Rankin Scale (mRS) (Note: mRS range: 0 (no residual symptoms) to 6 (death)

SECONDARY OUTCOMES:
Disability-weighted (or utility-weighted) mRS | 90 (±14) days after treatment initiation
  Standard utility weights applied to the mRS categories as follows: 1.0 for mRS level 0; 0.91 for mRS level 1; 0.76 for mRS level 2; 0.65 for mRS level 3; 0.33 for mRS level 4; 0 for mRS level 5; and 0 for mRS level 6
Return to the pre-stroke mRS level | 90 (±14) days after treatment initiation
  Returning to the pre-stroke mRS level post stroke
EQ-5D-5L | 90 (±14) days after treatment initiation
  Quality of life assessment scale with range: 0 (worst health) to 100 (best health)
Academic Medical Center - Linear Disability Scale (ALDS) | 90 (±14) days after treatment initiation
  Generic item bank that measures the disability status of patients with a broad range of diseases, as expressed by the ability to perform activities in daily living.

OTHER OUTCOMES:
modified Rankin Scale (mRS) | At hospital discharge
  Score of 0-3, 4, 5 or 6 on the modified Rankin Scale (mRS) (Note: mRS range: 0 (no residual symptoms) to 6 (death)
Montreal Cognitive Assessment (MoCA) | 90 (±14) days after treatment initiation
  Montreal Cognitive Assessment (MoCA) (Note: MoCA range: 0-30, higher scores mean better outcome)
Barthel Index Scale | 90 (±14) days after treatment initiation
  Barthel Index range: 0-100, higher scores mean participant is independent
Initial residence level or better time during first 90 days post-stroke | 90 days after treatment initiation
  Number of days spend at the initial residence level or better during the first 90 days post-stroke
Zarit's Burden Interview (ZBI) | 90 (±14) days after treatment initiation
  ZBI is a measure of caregiving burden that includes a 22 item interview. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). We will use the 4 item version of the ZBI which has good correlation with the full version.
Extended Thrombolysis in Cerebral Ischemia scale | At the end of EVT procedure
  The 7-point scale of eTICI is as follows: eTICI0 = 0% reperfusion; eTICI 1 = minimal flow past the occlusion but no perfusion ; eTICI2a = 1-49% reperfusion; eTICI2b50 = 50-66% reperfusion; eTICI2b67 = 67-89% reperfusion; eTICI2c = 90-99% reperfusion; eTICI3 = complete reperfusion
Death | 90 (±14) after treatment initiation
Symptomatic intracranial hemorrhage | 24 (±6) hours
  Evaluate modified Heidelberg definition

CONTACTS AND LOCATIONS:
Overall Officials: Eva Mistry, MD, Principal Investigator — University of Cincinnati; Jeffrey Saver, MD, Principal Investigator — Ronald Reagan UCLA Medical Center; J Mocco, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Heidi Sucharew, PhD, Principal Investigator — University of Cincinnati
Locations (19):
- United States (19):
  - HonorHealth, Phoenix, Arizona
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University of California at Los Angeles, Los Angeles, California
  - Swedish Medical Center, Englewood, Colorado
  - Hartford Health Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas at Austin, Austin, Texas
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after completing of the final analysis